CLINICAL TRIAL: NCT01425112
Title: Clinical Trial Comparing Subconjunctival and Topical Bevacizumab as Adjuncts to Trabeculectomy in Improving Outcomes for Primary Open Angle Glaucoma
Brief Title: Comparison of Subconjuctival Versus Topical Bevacizumab as Adjunct Therapy to Trabeculectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sudhalkar Eye Hospital (Other)
Responsible Party: Principal Investigator, Aditya Sudhalkar, Dr. Aditya Anand Sudhalkar, Sudhalkar Eye Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 31234EH
Record Dates: First submitted 2011-08-25; First posted 2011-08-29 (Estimated); Last update posted 2011-08-29 (Estimated); Status verified 2011-08

CONDITIONS: Complications of Treatment; Progression
Keywords: trabeculectomy; bevacizumab; anti-VEGF; Efficacy
MeSH Terms: conditions — Disease Progression | interventions — Phacoemulsification

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Topical/Subconjunctival (Experimental): Depending upon the mode of administration
  Interventions: Procedure: Phacoemulsification

INTERVENTIONS:
Procedure: Phacoemulsification — Surgery for complications of trabeculectomy

SUMMARY:
Bevacizumab is an anti vascular endothelial growth factor(anti-VEGF) substance that is known to reduce neovascularization and fibrovascular proliferation in inflammatory conditions, including post-operative inflammation. It has shown efficacy in numerous ocular conditions(off-label), that includes Age related macular degeneration, proliferative diabetic retinopathy, neovascular glaucoma and corneal neovascularization. It is being explored as an option for preventing recurrence of pterygium and as an adjunct to improving outcomes of trabeculectomy. There is a debate as to the mode and duration of bevacizumab administration for trabeculectomy. This study aims to compare a single subconjunctival dose of bevacizumab with topical therapy over one month in terms of outcomes of trabeculectomy surgery, non-progression of field loss and stable intraocular pressure(IOP) control.

ELIGIBILITY:
Inclusion Criteria:

* Primary Open Angle Glaucoma
* Progression
* Failure to reach target IOP
* Non compliant

Exclusion Criteria:

* Resurgery
* Systemic contraindication to bevacizumab
* All other forms of glaucoma

Min Age: 42 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2007-12; Primary Completion 2011-05 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Intraocular pressure control | For 2 years

SECONDARY OUTCOMES:
Progression | 2 years